CLINICAL TRIAL: NCT06485830
Title: Effect of Neural Mobilization, Compared to Conventional Physical Therapy, in Children Diagnosed with Cerebral Palsy. a Pragmatic Approach
Brief Title: Neural Mobilization and Cerebral Palsy
Acronym: NEUROREHAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: Instituto de Biomedicina (IBiS) de Sevilla (Unknown)
Responsible Party: Principal Investigator, Alberto Marcos Heredia-Rizo, University Full Professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEUROREHAB
Record Dates: First submitted 2024-06-18; First posted 2024-07-03 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy; Neurologic Disorder
Keywords: range of motion; pain intensity; gross motor function; neural mobilisation; quality of life; muscle stiffness; muscle tension
MeSH Terms: conditions — Cerebral Palsy; Nervous System Diseases; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Sealed opaque envelopes will be used for treatment allocation. The research in charge of collecting the outcome measures will remained unaware of treatment allocation group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neural mobilization of the lower limb (Experimental): Several neural mobilization techniques will be performed for the lower limb, with a special focus on the sciatic nerve. First, three different passive techniques will be used. These will consist of two sets of ten repetitions each with one minute rest between sets. This will last approximately 5 minutes. Then, three dynamic neural mobilization techniques will be performed, with each exercise lasting for 5 minutes per set, including two different sets (one minute rest between them), with a total of 10 minutes of mobilization and one minute of rest per exercise. Therefore the complete approach will last for 30 minutes approximately. Following this set of dynamic neural mobilization exercises, static neural mobilizations of the sciatic nerve will be performed again following the same order and duration than in the beginning.
  Interventions: Procedure: Neural mobilization of the lower limb
- Conventional physiotherapy treatment (Active Comparator): A conventional treatment will be performed, consisting of passive and active mobilizations, active stretching, and techniques aimed at improving daily life activities
  Interventions: Procedure: Conventional physical therapy

INTERVENTIONS:
Procedure: Neural mobilization of the lower limb — Static neural mobilization techniques will be performed for the lower limb. Static procedures will consist of two sets of 10 repetitions, with one minute rest between sets. Next, dynamic neural mobilization techniques will be performed, with each exercise lasting 5 minutes per set, with one minute rest between them. Therefore, dynamic procedures will consist of 10 minutes per mobilization technique (with one minute rest between exercises).
  At the end of all dynamic mobilization exercises, static mobilizations of the sciatic nerve will be performed again in the same order and with the same duration.
  The intervention will consist of a total of 8 sessions (either twice a week for four weeks or once a week for a total of 8 weeks). This will depend on the participant usual attendance to his/her treatment center
  Other Names: Neurodynamics
  Arms: Neural mobilization of the lower limb
Procedure: Conventional physical therapy — The intervention will include a first part in which active mobilizations, active-assisted mobilizations, and active stretches will be performed, followed by activities aimed at improving physical training, mobility training, and strength training oriented towards specific tasks. After this second part, the first part will be repeated in the same order and duration.
  The intervention will consist of a total of 8 sessions (either twice a week for four weeks or once a week for a total of 8 weeks). This will depend on the participant usual attendance to his/her treatment center
  Other Names: Usual care
  Arms: Conventional physiotherapy treatment

SUMMARY:
Objective: To assess the effect of neural mobilization applied to the lower limbs, compared to conventional physical therapy, in children diagnosed with Cerebral Palsy. Using the International Classification of Functioning, Disability and Health, the investigators will try to evaluate the impact of the intervention in aspects related with structure, activity, and participation.This project will mainly focus on the structure dimension. More specifically, the investigators aim to observe if a treatment protocol designed to modify the structure (e.g.,the sciatic nerve using neural mobilization techniques), will evoke changes not only in the structural dimension, but also will be able to modify the activity and participation dimensions.

Design: A single blinded randomized clinical trial (the evaluator will remain blinded to treatment allocation group) will be conducted. The experimental group will receive an intervention consisting on the use of neurodynamic mobilization procedures of the lower limb and participants in the control group will undergo a conventional physical therapy intervention (stretching, mobilization), without the use of neural mobilization.

Subjects: Participants will be aged between 5 and 18 years, and with a confirmed diagnosed of Cerebral Palsy with the presence of spasticity in the lower limbs.

Methods: Participants will be randomly allocated into two groups: experimental or control group. The primary outcome will be the range of motion (flexion and extension) of the hip, knee and ankle. Secondary outcomes will include gross motor function, pain intensity, muscle stiffness, muscle tension, and functional measures.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents diagnosed with Cerebral Palsy or presence of spasticity and aged between 5 and 18 years.
* Level I to V in the Gross Motor Function Classification System, which denotes that the participant should be able to walk with or without using assistive devices.
* Increased muscle tone in the lower extremities, represented by a score greater than 0 on the Tardieu clinical scale and a positive response in the Duncan Ely test.
* Ability to communicate pain.
* Ability to follow simple commands.

Exclusion Criteria:

* Have ankle joint arthrodesis or any surgical operation that prevents joint mobilization of the lower limb to some degree.
* Any significant change in medication treatment during the study period that may influence (increase or decrease) muscle tone.
* Experience uncontrolled epileptic seizures despite medication.
* Have received botulinum toxin treatment in the lower limb within the 6 months prior to the study.
* Undergo a different physical therapy treatment parallel to that developed in the study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Range of motion | From baseline to up to 8 weeks, with a 3-month and a 6-month follow up
  Passive range of motion will be assessed for flexion and extension of the hip, knee, and ankle. Using a handheld goniometer, each joint will be measured three times, using the average of the three measures for subsequent analysis.

SECONDARY OUTCOMES:
Self-reported pain intensity | From Baseline to up to 8 weeks, with a 3-month and a 6- month follow up
  Current self-reported pain intensity during the most passive Straight Leg Rise test, as assessed with a 0 to 10 Numeric Pain Rating Scale (NPRS).T he Numeric Pain Rating Scale is a 11-point rating scale that ranges from 0, which denotes no pain at all, to 10, which denotes the maximum bearable pain. This has been selected as the most recommended and valid tool to evaluate self-reported pain intensity.
Spasticity | From Baseline to up to 8 weeks, with a 3-month and a 6- month follow up
  Spasticity of the hamstrings and adductor muscles will be measured using the modified Tardieu scale. The modified Tardieu Scale is the most common tool used in the clinical setting to evaluate the level of muscle spasticity. The muscle response to a slow and fast stretching will be collected. There are two parts to the assessment that are applied to each muscle group that is examined. In the first part of the assessment, the health professional slowly moves the person's limb to observe the full range of their available movement. In the second part of the assessment, the same limb is moved quickly. Both range of motions (in response to a slow and a fast movement) will be measured using a goniometer. Higher scores represent a lower level of spasticity
Activity and Participation | From Baseline to up to 8 weeks.,with a 3-month and a 6- month follow up
  The Gross Motor Function Classification System will be used to assess activity dimensions related to standing and walking, while the Functional Mobility Scale will evaluate participation by measuring the time taken to walk 5 and 50 meters. Final scores in the Gross Motor Function Classification System will be categorised in five different levels (I to V), with lover levels denoting higher level of walking independence. For the Functional Mobility Scale, a rating of 1, 2, 3, 4, 5 or 6 is given for each distance, with higher values representing higher levels of independence.
Health-related quality of life | From Baseline to up to 8 weeks, with a 3-month and a 6- month follow up
  The Cerebral Palsy Quality of Life Questionnaire will be given to parents or legal tutors of participants (when applicable) or to study participants (depending on their age) to analyze the relationship of the condition with the environment. There are different versions, including a primary caregiver/parent report for children aged 4 to 12 years; and a self-report for children aged 9 to 12 years. Another version has been designed for adolescents aged 13-18 years. Higher scores denote higher levels of well-being.
Myotonometry | From Baseline to up to 8 weeks, with a 3-month and a 6- month follow up
  Muscle tone and muscle stiffness will be measured using a myotonometer. Assessment points will be marked with a non-invasive demographic pencil on the select points: hamstring muscles, the rectus femoris muscle, and the adductor muscle. Two points will be located in the muscle belly of the abovementioned muscles. At each point, muscle tone and stiffness will be measured using a device called MyotonPRO MyotonPRO (Myoton AS, Estonia). The MyotonPRO is small,non-invasive, and it has shown good validity and high reliability in larger and smaller body muscles.This device delivers a multi-scan mode of three brief mechanical impulses, each one shortly followed by a quick release, to record the damped natural oscillation of the muscle using an accelerometer. Evaluations will be made in both sides.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto M. Heredia Rizo, PhD, Study Director — Instituto de Biomedicina (IBiS) de Sevilla
Locations (2):
- Spain (2):
  - Centro de Atencion Infantil Temprana (CAIT), Universidad de Cordoba, Córdoba, Cordoba
  - University of Sevilla, Seville, Sevilla

IPD SHARING:
Plan to Share IPD: Yes
Individual participation data will be made available in the repository of the University of Seville, Spain
Supporting Information: ICF, CSR
Time Frame: Data will become available once the study has been published with no limit for accessibility.
URL: https://idus.us.es/